CLINICAL TRIAL: NCT06790446
Title: Plantar-flexor Structural and Neural Changes in Chronic Hemiparesis Following Two Months of Eccentric Training: a Pilot, Randomized Controlled Trial
Brief Title: Plantar Flexor Eccentric Training in Chronic Hemiparesis
Acronym: EXC-AVC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuroloco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-061; 2021-A01201-40 (Other: Hôpitaux Universitaires Henri Mondor)
Record Dates: First submitted 2025-01-14; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Hemiparesis
Keywords: Spastic myopathy; Eccentric training; Plantar flexors; Spastic cocontraction; Paresis
MeSH Terms: conditions — Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eccentric training group (ECC) (Experimental): In this group, participants come three times a week during 8 weeks at the Henri Mondor University Hospital to complete their isokinetic eccentric training sessions
  Interventions: Other: Eccentric training group (ECC)
- Conventional therapy group (Active Comparator): In this group, participants continue on the routine community-based therapy carried out in private practice or at home. Quantitative and qualitative description of this rehabilitation will be collected using questionnaires at the end of the experimental phase
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Other: Eccentric training group (ECC) — The first, preparatory phase, lasts two weeks, aiming at making the participant familiar with the principles of eccentric training. Participants first experience the muscle recruitment patterns (during two sessions), then are prepared to induce protective response from the plantar flexors, conditioning these muscles for higher subsequent eccentric intensities.
  The aim of the second, training phase per se, which lasts six weeks, is to induce muscular and neurological adaptations through a steady increase in work intensity to stimulate muscle plasticity until the end of the program - varying volume, load and speed.
  Perceived exertion is quantified using Borg's scale (expected rating between 3 and 6) to ensure sufficient work intensity and prevent excessive fatigue. Musculoskeletal pain is assessed before and after each session through a Visual Analog Scale (0-10). Verbal encouragements and advising on correct exercise execution are provided by the therapist along each session.
  Arms: Eccentric training group (ECC)
Other: Conventional therapy — The participant visits a physiotherapist depending on the prescription, as in current practice
  Arms: Conventional therapy group

SUMMARY:
The goal of this clinical trial is to assess the effects of a plantar flexor eccentric training on muscle health of these muscles and teir descending command in chronic spastic hemiparesis. The effects of the strength and lower limb function will also be explored.

The main question of this study is : do MG and SOL fascicle length and thickness can be modified after 2-months of eccentric training ? The experimental treatment will be compared to conventional therapy group (Gold standard).

At D1, participants will be randomized into 2 groups: eccentric training versus conventional therapy for 8-weeks. Every participant will be assessed by blinded investigators at D1 and W8.

In the eccentric training, patients will receive 3 sessions/week of a customized isokinetic eccentric program. in the control group, patients will follow their sessions of rehabilitation as before their inclusion.

DETAILED DESCRIPTION:
Background: Functional deficits in stroke patients with hemiparesis result from muscular damage, known as spastic myopathy, and neurological damage, combining agonist paresis and antagonist hyperactivity. In the chronic phase, it has been shown that conventional rehabilitation does not improve function beyond an average 0.04 m/sec increase in walking speed in hemiparesis patients. On the other hand, eccentric exercise has been shown in healthy subjects to markedly improve muscle extensibility, neuronal efficiency and muscle strength. However, its effects on spastic muscles in the chronic post-stroke phase, and in particular on plantar flexors, remain poorly documented and contradictory. Such an intervention, targeting the plantar flexor muscles of the subjects, could act both on spastic myopathy by reducing passive stiffness and increasing length and thickness, but also on propulsion capacity in walking, thus improving their walking speed.

Primary objective: To evaluate the effect on plantar flexor architectural parameters of an isokinetic eccentric exercise protocol targeting these muscles compared with conventional rehabilitation.

Secondary objectives: To compare each of the changes in the secondary endpoints in subjects with chronic post-stroke hemiparesis after 8 weeks of a plantar flexor eccentric exercise program compared with conventional rehabilitation (W8-D1).

Participants: 20 subjects with hemiparesis will be recruited and randomly assigned to 2 groups: eccentric training (ECC) versus conventional rehabilitation (CONV) Inclusion criteria are (a) adults aged 18 to 80 years, (b) chronic hemiparesis (> 6 months), (c) walking speed > 0.2 m/sec, unassisted over 10m, (d) stable hemiparesis with plantar flexor involvement, (e) written consent.

Intervention: The plantar flexor eccentric training group will carry out its sessions on an isokinetic dynamometer (Contrex) at a rate of 3 sessions per week for 8 weeks. Each session will consist of a warm-up (10 concentric plantar flexions at 30°/s). The rehabilitation protocol will be carried out in 2 parts. The first 2 weeks will be a period of familiarization and adaptation to the contraction mode, to minimize risks and optimize tissue adaptations. Then, during the following 6 weeks, the intensity of the exercises will gradually increase, modifying the speed, the load and the volume (number of repetitions). Quantification of the subject's load and pain status will be assessed using the force curves of the isokinetic dynamometer and a visual analog scale, respectively.

Outcome measures: Assessments will be made at the first and last sessions. The primary outcome will be the structural changes (fascicular length and thickness) of medial gastrocnemius and soleus (through ultrasound). Secondary endpoints will be , biomechanical (change in peak isometric force of plantar flexors during maximal voluntary contraction, neurophysiological (changes in the agonist and the antagonist activation of the medial gastrocnemius and soleus, and functional (change in maximum barefoot walking speed over 10m (AT10)). Also, correlations between change in gait speed and change in fascicular length of the medial gastrocnemius and soleus on the paretic side, as well as between change in gait speed and change in peak force of the paretic plantar flexors will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* adults with chronic hemiparesis (> 6 months)
* XV1-GAS<100°
* walking speed > 0.2 m/sec
* unassisted over 10m
* stable hemiparesis with plantar flexor involvement
* written consent

Exclusion Criteria:

* cognitive impairment (MoCa<26),
* orthopedic or traumatic ankle involvement,
* medical contraindication to maximal effort,
* follow-up of another research program,
* sural triceps toxin injection < 3 months,
* adjacent neurological pathology,
* pregnant women,
* women of childbearing age who are not on effective contraception, either mechanical (IUD) or hormonal (pill),
* wearing a pacemaker or implanted defibrillator,
* persistent cardiovascular disorders following a cardiac accident,
* wearing an implanted medical device
* a history of epilepsy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-02-27 (Actual); Study Completion 2022-02-27 (Actual)

PRIMARY OUTCOMES:
MG and SOL Architectural parameters | Day 0 ; Month 2
  To quantify thickness and fascicle length (Lƒ) of soleus, then of medial gastrocnemius, participants were seated in the isokinetic ergometer: hip flexion at 45°, paretic knee extended, and the paretic ankle positioned at 80% of XV1-GAS (i.e. 80% of maximal clinical extensibility of the gastro-soleus complex). Three ultrasound images for each muscle are collected under passive conditions. Prior detection of skin landmarks allows standardization of the probe location. For collection of MG muscle images, the probe is positioned midway along the muscle body. For SOL, the probe is placed directly below the MTJ-MG.

SECONDARY OUTCOMES:
peaktorque in dorsiflexion / plantarflexion | Day 0 ; Month 2
  Following the collection of ultrasound images, the subject in the ergometer was asked to perform isometric Maximal Voluntary Contraction (MVC) into plantar flexion, then into dorsiflexion, through three consecutive trials at a 90° position of XV1-GAS (ankle at 90°). Each measurement is applied in a standardized manner including a warm-up effort before the first trial, one maximal effort to be held for five seconds, and two minutes of rest before the next trial. The best of the three peak torque measurements is collected
MG and SOL Coefficients of agonist activation and antagonist activation | Day 0 ; Month 2
  EMG activities of soleus and gastrocnemius are recorded during each trial of isometric Maximal Voluntary Contraction (MVC) into plantar flexion, and into dorsiflexion.
  Coefficients of AGonist activation (CAG-SO, CAG-MG) and of ANtagonist activation (CAN-SO, CAN-MG) during maximal voluntary efforts are calculated for MG and SOL muscles. CAG-MG and CAG-SOL are defined as the ratio between the RMS-EMG of the maximal activity of the muscle during MVC over its Mmax obtained through supramaximal neurostimulation, using a classic technique of incremental stimulations until no more increase in the M response occurs. Coefficients of ANtagonist activation CAN-SO, CAN-MG are quantified as the ratio of the RMS (500 ms) of the muscle EMG activity during maximal dorsiflexion (co-activation) over its Mmax. Importantly, the Mmax obtained at baseline (Day 0) is kept as the reference for a given muscle throughout measurements, whether at Day 0 or Month 2.
Ambulation speed | Day 0 ; Month 2
  Maximal barefoot ambulation speed is measured over ten meters without technical aid, following the conditions of the AT10 (10-meter Ambulation Test) with start and end seated

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires Henri Mondor, Créteil, Île-de-France Region, France